CLINICAL TRIAL: NCT03587103
Title: Learning Implementation of Guideline-based Decision Support System for Hypertension Treatment: Testing Alternative Antihypertensive Regimens Using ACE-Inhibitors, Calcium Channel Blockers and Diuretics (LIGHT-ACD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-I2M-1-006-2
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Fumigant 93

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Protocol initiate with A (Experimental): Eligible participants will be randomized to receive one of the protocols initiated with A, or the protocols initiated with two-drug combination therapy with full dose A.
  Interventions: Behavioral: Protocol initiate with A
- Protocol initiate with C (Experimental): Eligible participants will be randomized to receive one of the protocols initiated with C, or the protocols initiated with two-drug combination therapy with full dose C.
  Interventions: Behavioral: Protocol initiate with C
- Protocol initiate with D (Experimental): Eligible participants will be randomized to receive one of the protocols initiated with D, or the protocols initiated with two-drug combination therapy with full dose D.
  Interventions: Behavioral: Protocol initiate with D

INTERVENTIONS:
Behavioral: Protocol initiate with A — The BP-lowering medication adjustment and titration will follow A-AC-ACD or A-AD-ADC for individuals randomized to A or two-drug combination therapy with full dose of A in their initial medication assignment.
  Arms: Protocol initiate with A
Behavioral: Protocol initiate with C — The BP-lowering medication adjustment and titration will follow C-CA-CAD or C-CD-CDA for individuals randomized to C or two-drug combination therapy with full dose of C in their initial medication assignment.
  Arms: Protocol initiate with C
Behavioral: Protocol initiate with D — The BP-lowering medication adjustment and titration will follow D-DA-DAC or D-DC-DCA for individuals randomized to D or two-drug combination therapy with full dose of D in their initial medication assignment.
  Arms: Protocol initiate with D

SUMMARY:
This trial aims to compare the efficacy of several guideline-based hypertensive medication regimens initiated with Angiotensin Converting Enzyme Inhibitor/Angiotensin Receptor Blocker [A], Calcium Channel Blocker [C] and Diuretic [D].

DETAILED DESCRIPTION:
The LIGHT-ACD Trial is conducted based on the LIGHT trial and aims to compare the efficacy of several guideline-based hypertensive medication regimens initiated with A, C and D for BP control.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥18 years
2. Local resident of the community/township who attend a PHC center with DSS treatment of hypertension
3. Established diagnosis of essential hypertension, with SBP≥140mmHg and <180mmHg
4. Not currently taking any antihypertensive medication or taking only one antihypertensive medication which in not B

Exclusion criteria:

1. History of coronary heart disease (i.e., angina, MI, CABG, PCI, >50% stenosis of coronary artery, or positive stress test)
2. Physician-diagnosed or self-reported CKD, eGFR <60 mL/min/1.73m2 (if serum creatinine available), or currently on dialysis
3. Physician-diagnosed diabetes mellitus
4. Physician-diagnosed heart failure
5. Physician-diagnosed secondary hypertension
6. Intolerance to any class of antihypertensive medications among A, C or D
7. Other serious medical illness such as malignant cancer, hepatic dysfunction, et al.
8. Currently at the acute phase of any diseases
9. Subject is pregnant or breast feeding, or planning to become pregnant or breast feeding during study period
10. Patients measured blood pressure at home and the average self-measured home blood pressure <135/85mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2019-08-21 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Average change in BP from first visit after the decision support system is installed to 9-month among the individuals who initiated with A, C, and D (population 1) and among those who initiated with two-drug therapy with AC, AD or CD (population 2) | Baseline; 1 year
  Average change in BP from first visit after the decision support system is installed to 9-month among population 1 (SBP 140-159 mmHg, not currently taking any antihypertensive medications) who initiated with A, C, and D and among population 2 (SBP≥160 mmHg, taking 0-1 antihypertensive medications which is not B; or SBP 140-159mmHg, taking one antihypertensive medication which is not B) who initiated with two-drug therapy with AC, AD or CD, respectively.

SECONDARY OUTCOMES:
Proportion of individuals with BP<140/90 mmHg at 9 month. | Baseline; 1 year
  Proportion of individuals with BP<140/90 mmHg at 9 month among the individuals (population 1: SBP 140-159 mmHg, not currently taking any antihypertensive medications) who initiated with A, C, and D, among those (population 2: SBP≥160 mmHg, taking 0-1 antihypertensive medications which is not B; or SBP 140-159mmHg, taking one antihypertensive medication which is not B) who initiated with two-drug therapy with AC, AD or CD.
Proportion of individuals with BP<160/100 mmHg at 9 month. | Baseline; 1 year
  Proportion of individuals with BP<160/100 mmHg at 9 month among the individuals (population 1: SBP 140-159 mmHg, not currently taking any antihypertensive medications) who initiated with A, C, and D, among those (population 2: SBP≥160 mmHg, taking 0-1 antihypertensive medications which is not B; or SBP 140-159mmHg, taking one antihypertensive medication which is not B) who initiated with two-drug therapy with AC, AD or CD separately.
Proportion of individuals who received monotherapy, two-drug treatment, three-drug treatment, or referral at 9 month. | Baseline; 1 year
  Proportion of individuals who received monotherapy (only in populations 1), two-drug treatment, three-drug treatment, or referral at 9 month among the individuals (population 1: SBP 140-159 mmHg, not currently taking any antihypertensive medications) who initiated with A, C, and D, among those (population 2: SBP≥160 mmHg, taking 0-1 antihypertensive medications which is not B; or SBP 140-159mmHg, taking one antihypertensive medication which is not B) who initiated with two-drug therapy with AC, AD or CD.
Proportion of individuals intolerant to each of the four medications. | Baseline; 1 year
  Proportion of individuals intolerant to each of the four medications among the individuals (population 1: SBP 140-159 mmHg, not currently taking any antihypertensive medications) who initiated with A, C, and D, among those (population 2: SBP≥160 mmHg, taking 0-1 antihypertensive medications which is not B; or SBP 140-159mmHg, taking one antihypertensive medication which is not B) who initiated with two-drug therapy with AC, AD or CD.
Proportion of individuals who switched to usual care for any reason. | Baseline; 1 year
  Proportion of individuals who switched to usual care for any reason among the individuals (population 1: SBP 140-159 mmHg, not currently taking any antihypertensive medications) who initiated with A, C, and D, among those (population 2: SBP≥160 mmHg, taking 0-1 antihypertensive medications which is not B; or SBP 140-159mmHg, taking one antihypertensive medication which is not B) who initiated with two-drug therapy with AC, AD or CD.

OTHER OUTCOMES:
Comparison of average change in BP from the first visit after randomization to 9-month between A-AC-ACD and A-AD-ADC, C-CA-CAD and C-CD-CDA, and D-DA-DAC or D-DC-DCA only in population 1, respectively. | Baseline; 1 year
  Comparison of average change in BP from first visit after randomization to 9-month between protocol A-AC-ACD and A-AD-ADC, C-CA-CAD and C-CD-CDA, and D-DA-DAC or D-DC-DCA among population 1(SBP 140-159 mmHg, not currently taking any antihypertensive medications) .

CONTACTS AND LOCATIONS:
Overall Officials: Xin Zheng, MD, PhD, Principal Investigator — China National Center for Cardiovascular Disease
Locations (3):
- China (3):
  - Luoyang Oriental hospital, Beijing, Henan
  - Yankuang Hospital, Zoucheng, Shandong
  - Center for chronic disease control, Shenzhen, ShenZhen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Song J, Wang X, Wang B, Gao Y, Liu J, Zhang H, Li X, Li J, Wang JG, Cai J, Herrin J, Armitage J, Krumholz HM, Zheng X; LIGHT Collaborative Group. Effectiveness of a clinical decision support system for hypertension management in primary care: study protocol for a pragmatic cluster-randomized controlled trial. Trials. 2022 May 16;23(1):412. doi: 10.1186/s13063-022-06374-x. PMID 35578345